CLINICAL TRIAL: NCT05417061
Title: Serum and Saliva Sirtuin 6, Lipoxin A4, Caspase8 Levels in Correlation With Periodontal Status in Severe Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nur Balci, DDs, PhD, ASSOC. PROF DR, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 138
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-06

CONDITIONS: Periodontitis; Diagnose Disease
Keywords: inflammation resolution; periodontitis; cell apoptosis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Saliva and serum of periodontitis patients collected for analyzing SIRT6, LPXA4, CASP8
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saliva and serum collection of patients and samples molecules analysis (Active Comparator)
  Interventions: Other: Saliva and serum sampling
- Salivary and serum SIRT6, LPXA4 and CASP8 observation (Experimental): Saliva and serum samples obtained for each patient were used for cytokine analysis. Prepared samples were analyzed for Lipoxin A4 (LXA4), Caspase 8 (CASP8) and Sirtuin-6 (SIRT6) using commercial ELISA kits
  (Elabscience, Houston, Texas, USA and Bioaasay Technology Laboratory (BT-Lab), Shanghai, China, respectively) according to the manufacturer's instructions. The detection limits of ELISA kits were 0.78 - 50ng/ml for LXA4, 0.16 - 10ng/ml for CASP8 and 0.1- 40 ng/ml for SIRT6.
  Interventions: Other: Saliva and serum sampling

INTERVENTIONS:
Other: Saliva and serum sampling — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes.
  Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff (MFD) from each participant. Saliva and serum were then stored at -80 °C until analysis.

SUMMARY:
It has been stated that Sirtuin-6 (SIRT6) play a important role in regulation of inflammation, energy metabolism, homeostasis and apoptosis, and SIRT6 may be assosiciated with many diseases. The aim of this study was to evaluate saliva and serum SIRT6, Lipoxin A4 (LXA4) and Caspase-8 (CASP8) levels in correlation with periodontal clinical status in patients with periodontitis and healthy subjects

DETAILED DESCRIPTION:
20 patients with Stage III Grade B periodontitis (P) and 20 periodontally healthy individuals (control;C) were included in this study. Clinical periodontal parameters were measured. Saliva and serum levels of SIRT6, LXA4 and CASP8 were analyzed by enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* clinical diagnosis of periodontitis
* clinical diagnosis of periodontal health

Exclusion Criteria:

* history of regular use of systemic antibiotics anti-inflammatory, or antioxidant drugs (previous 3 months)
* nonsurgical periodontal treatment (previous 6 months)
* surgical periodontal treatment (previous 12 months)
* presence of<10 teeth
* current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy)
* diabetes
* diagnosis of rheumatoid arthritis
* pregnancy
* lactating
* smoking
* excessive alcohol consumption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | 6 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
Clinical attachment level | 6 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
Bleeding on probing | 6 months
  referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth.

SECONDARY OUTCOMES:
Saliva and serum samples processing and analyses | 2 months
  Saliva and serum samples obtained for each patient were used for cytokine analysis. Prepared samples were analyzed for Lipoxin A4 (LXA4), Caspase 8 (CASP8) and Sirtuin-6 (SIRT6) using commercial ELISA kits
  (Elabscience, Houston, Texas, USA and Bioaasay Technology Laboratory (BT-Lab), Shanghai, China, respectively) according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cekici A, Sahinkaya S, Donmez MF, Turkmen E, Balci N, Toygar H. Sirtuin6 and Lipoxin A4 levels are decreased in severe periodontitis. Clin Oral Investig. 2023 Dec;27(12):7407-7415. doi: 10.1007/s00784-023-05330-6. Epub 2023 Oct 18. PMID 37851128